CLINICAL TRIAL: NCT04106882
Title: Dynamic Connectivity Under Metabolic Constraints
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: Martinos Center for Biomedical Imaging (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017D001434
Record Dates: First submitted 2019-09-17; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Insulin Resistance; Healthy; Diet Modification; Aging
Keywords: insulin resistance; exogenous ketone; glucose; diet; aging
MeSH Terms: conditions — Insulin Resistance | interventions — Ketones; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Metabolic Manipulation via Diet fMRI (Experimental): All subjects are tested three times, each in a different diet-induced metabolic state: glycolytic (glucose burning), fasting (8 hours no food), and ketotic (fat burning). While having their brains scanned with MRI, subjects are initially tested at rest, and then perform a task. Midway through the session, subjects are removed from the scanner and drink up to 75g glucose. Data analyses quantify network reorganization in response to changing energy constraints (i.e., cognitive demand, fuel).
  Interventions: Drug: Glucose
- Arm 2: Metabolic Manipulation via Ketone Supplement fMRI (Experimental): All subjects are tested twice, both times in a fasting condition (8 hours no food, unrestricted water). While having their brains scanned with MRI, subjects are initially tested at rest, and then perform a task. Midway through the session, subjects are removed from the scanner and drink either of two fuel sources. In the ketotic (ketone burning) session they will drink a ketone sports drink dosed at 395mg/kg. During the glycolytic (glucose burning) session the same subjects will drink a bolus of glucose, calorie-matched to the ketones. Data analyses quantify network reorganization in response to changing energy constraints (i.e., cognitive demand, fuel).
  Interventions: Drug: Ketones; Drug: Glucose
- Arm 3: Metabolic Manipulation via Ketone Supplement MR/PET (Experimental): All subjects are tested twice, both times in a fasting condition (8 hours no food, unrestricted water). For both sessions, the investigators will intravenously administer the FDG radioisotope continuously throughout the scan. Thus, PET will map glucose uptake across the brain, while MRS is simultaneously used to measure production of the neurotransmitters glutamine and GABA. While having their brains scanned with MR/PET, subjects are initially tested at rest, and then perform a task. Subjects will drink a ketone sports drink dosed at 395mg/kg. During the glycolytic (glucose burning) session the same subjects will drink a bolus of glucose, calorie-matched to the ketones.
  Interventions: Drug: Ketones; Drug: Glucose

INTERVENTIONS:
Drug: Ketones — Supplement administered mid-scan.
  Arms: Arm 2: Metabolic Manipulation via Ketone Supplement fMRI; Arm 3: Metabolic Manipulation via Ketone Supplement MR/PET
Drug: Glucose — Supplement administered mid-scan.

SUMMARY:
The investigators are studying the impact of insulin resistance on the acceleration of brain aging and testing whether increased neuron insulin resistance can be counteracted by utilization of alternate metabolic pathways (e.g., ketones rather than glucose). This study has three Arms, which together provide synergistic data. For all three Arms, subjects are tested in a within-subjects design that consists of 2-3 testing sessions, 1-14 days apart, and counter-balanced for order. Impact of fuel (glucose in one session, ketones in the other) on brain metabolism and associated functioning is measured during each session. For Arms 1-2, the primary experimental measure is functional magnetic resonance imaging (fMRI), which is used to trace the self-organization of functional networks following changes in energy supply and demand. Arm 1 tests the impact of endogenous ketones produced by switching to a low carbohydrate diet, while Arm 2 tests the impact of exogenous ketones consumed as a nutritional supplement. For Arm 3, simultaneous magnetic resonance spectroscopy/positron-emission tomography (MR/PET) is used to quantify the impact of exogenous ketones on production of glutamate and GABA, key neurotransmitters.

Subjects will be given the option to participate in more than one of the Arms, but doing so is not expected nor required.

Prior to scans, subjects will receive a clinician-administered History and Physical (H&P), which includes vital signs, an oral glucose tolerance test (OGTT), and the comprehensive metabolic blood panel. These will be used to assess diabetes, kidney disease, and electrolytes. If subjects pass screening, they will be provided the option to participate in one or more Arms, which include neuroimaging. To provide a quantitative measure of time-varying metabolic activity throughout the scan, based upon quantitative models of glucose and ketone regulation, as well as to be able to implement safety stopping rules (see below), the investigators will obtain pin-prick blood samples three times: prior to the scan, following consumption of the glucose or ketone drink, and following completion of the scan. To assess effects of increased metabolic demand, the investigators measure brain response to cognitive load, transitioning from resting-state to spatial reasoning through a spatial navigation video task. To assess effects of increased metabolic supply, the investigators measure brain response to glucose or ketone bolus.

ELIGIBILITY:
Exclusion Criteria:

* claustrophobia
* history of neurological disease, heart attack, stroke, kidney disease, or myxedema
* chronic usage of alcohol
* current usage of psychotropic medication
* Type 1 diabetes mellitus
* Regular consumption of insulin, Metformin® or other medications (statins, NSAIDs, beta-blockers, glucocorticoids) that affect glucose and/or insulin utilization.
* difficulty swallowing
* pregnancy
* breastfeeding
* For PET: research imaging-related radiation exposure that exceeds current MGH Radiology Radiation Safety Commitee guidelines.

Inclusion Criteria:

* BMI < 30
* MRI compatible
* For PET with Optional 150 ml Blood Sampling Only: Must weigh at least 110 lbs to minimize risks per PHRC guidelines.
* 20/20 vision or correctable to 20/20 with contact lenses

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-06-19 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Diet related changes in brain network stability will be assessed by fMRI BOLD measurements. | Within two weeks of enrollment completion
  Changes in BOLD signal measurements will be observed between baseline and during a glycolytic, fasting, or ketotic state.
Glucose uptake will be measured by PET, with and without ketone supplement | Within two weeks of enrollment completion
  Continuous FDG PET infusion is used as a measure of glucose uptake during rest and task, with and without the ketone supplement.
Neurotransmitter production with and without ketone supplement will be measured by magnetic resonance spectroscopy | Within two weeks of enrollment completion
  Changes in neurotransmitter concentration under metabolic demands (i.e., task vs resting-state) with and without ketone supplement will be assessed by magnetic resonance spectroscopy.

SECONDARY OUTCOMES:
Cognitive performance will be assessed by Mini Mental State Exam (MMSE). | Within two weeks of enrollment completion
  All subjects will undergo cognitive testing prior to MRI scanning using the MMSE exam.
Cognitive performance will be assessed by CNS Vital Signs. | Within two weeks of enrollment completion
  All subjects will undergo cognitive testing prior to MRI scanning using the CNS Vital Signs exam.
Insulin resistance will be assessed by HbA1C. | Within two weeks of enrollment completion
  All subjects will be tested for insulin resistance prior to MRI scanning using veinous blood collected and tested for HbA1C.
Insulin resistance will be assessed by blood insulin level. | Within two weeks of enrollment completion
  All subjects will be tested for insulin resistance prior to MRI scanning using veinous blood collected and tested for insulin during a 2-hour Oral Glucose Tolerance Test (OGTT).
Insulin resistance will be assessed by blood glucose level. | Within two weeks of enrollment completion
  All subjects will be tested for insulin resistance prior to MRI scanning using veinous blood collected and tested for glucose during a 2-hour Oral Glucose Tolerance Test (OGTT).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Martinos Center for Biomedical Research, Building 149, Charlestown, Massachusetts
  - Bioengineering Building , Stony Brook University, Stony Brook, New York